CLINICAL TRIAL: NCT02597959
Title: Exposure Assessment and Intervention for Reducing Musculoskeletal Stresses and Work-related Injuries Among Allied Health Professionals in Surgical Care
Brief Title: Reducing Musculoskeletal Stresses and Work-related Injuries Among Allied Health Professionals in Surgical Care
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Susan Hallbeck, Ph.D., Senior Associate Consultant II, Mayo Clinic
Other Study IDs: 15-002833
Record Dates: First submitted 2015-08-13; First posted 2015-11-05 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Musculoskeletal Injury; Musculoskeletal Illness
Keywords: ergonomic risk factors; allied health professionals; surgical care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- risk factors of musculoskeletal injuries: trainees for surgical assistants - determining the level of risk
- design wearable devices: Creating feedback mechanism to reduce surgical assistant musculoskeletal risk

SUMMARY:
1. What are the risk factors that contribute to musculoskeletal injuries and fatigue on allied health professionals in surgical care (e.g. scrub nurses, surgical assistants, and circulating nurses)?
2. Can the investigators design wearable devices that the investigators can later evaluate?

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Employed at Mayo Clinic Rochester as Surgical Assistant, Circulating Nurse, and Scrub Nurse (Surgical Technicians)

Exclusion Criteria, Aims 1 and 2:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Surgical Assistants, Circulating Nurses, and Scrub Nurses (Surgical Technicians) employed at Mayo Clinic Rochester, MN, are the subjects for Aims 1 and 2. The subject population for the future Aim 3 includes surgical assistant anatomy laboratory students enrolled through the Mayo School of Health Sciences Surgical First Assistant Program, fall 2015.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2015-09; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Frequency of awkward postures | 4 months
  Awkward postures will be quantified with motion tracking using an inertial measurement unit (IMU), a lightweight, small sensor. IMU data will be collected and transmitted wirelessly to a real time monitoring system.

SECONDARY OUTCOMES:
Open-ended questionnaire on workflow and usability process to develop automated, unobtrusive, and cost-effective wearable device | 3 months
  Description: Open-ended questionnaire will present participants with the following questions after viewing a presentation on surgical ergonomics and vibrotactile feedback: "Would this device interrupt your work; if so, in what ways," "Are you concerned you may be distracted," Might it interfere with movement in any way," "Could you provide feedback on the vibration settings," etc.time work postures and these data will control tactor activation.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hallbeck, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States